CLINICAL TRIAL: NCT00984451
Title: A Pilot Study for Collection of Anti-Influenza A Immune Plasma
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: 09-I-0226; 09-I-0226; IRC001
Record Dates: First submitted 2009-09-24; First posted 2009-09-25 (Estimated); Last update posted 2019-08-19 (Actual); Status verified 2019-08

CONDITIONS: Influenza A Virus Infection; Swine Flu
Keywords: Antibody Treatment; Immune Therapy; Infectious Diseases; IVIG; Plasma Apheresis; Influenza A; Swine Flu
MeSH Terms: conditions — Orthomyxoviridae Infections; Communicable Diseases | interventions — Vaccination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: Plasma collection following infection or vaccination with influenza A — High titer influenza A plasma collection for use as therapeutic plasma in influenza treatment studies.

SUMMARY:
Background:

* The influenza A virus can cause infections that lead to fever, cough, muscle aches, diarrhea, and headaches, and can even be fatal in some people. Seasonal influenza kills an estimated 36,000 people in the United States each year. In addition, more than 200,000 people are hospitalized for flu-related complications. Influenza A has a substantial health effect on every age group.
* Currently, treatments are available for influenza A, but there is concern that the rate of complications or even death from this infection is still high despite treatment, and that over time this virus may become resistant to these treatments. Researchers are interested in developing a possible new treatment that uses antibodies against influenza A virus.

Objectives:

- To collect plasma (the liquid component of blood containing antibodies) from people who have high levels of antibodies against the influenza A virus because they either have been previously infected with the virus or have been vaccinated against the infection.

Eligibility:

* Healthy male volunteers between 18 and 60 years of age who are eligible to donate blood.
* Individuals must have previously either recovered from influenza infection or have been vaccinated against the infection, and may be subject to other restrictions on participating in National Institutes of Health research studies.

Design:

* Volunteers will undergo apheresis, an outpatient procedure in which researchers will collect plasma containing antibodies against the influenza virus by drawing blood into a special machine that separates blood cells from the liquid portion under sterile conditions and then returns the blood cells to the donor.
* Volunteers will be screened with blood tests to ensure that they are eligible to participate and donate blood.
* Volunteers are asked to undergo at least 3 sessions of apheresis; if willing, they can volunteer to participate in up to 20 sessions.
* After plasma is collected, it will be tested to ensure that it can be used to safely develop treatments for patients who have influenza A infection.

DETAILED DESCRIPTION:
Two types of influenza A widely circulate in humans and cause seasonal outbreaks and epidemics - H1N1 (swine flu) and H3N2 (a subtype abundant in seasonal influenza). During the 2009-2010 influenza season, the most commonly reported virus was influenza A (H1N1). However, during the 2010-2011 influenza season, the most commonly reported virus was influenza A (H3N2), but influenza A (H1N1) viruses and influenza B viruses circulated as well.

A certain age group may be hit harder by one type of influenza virus than another (for example, the 2009 H1N1 virus disproportionately affected people younger than 65 years of age rather than those older than 65, whereas H3N2 virus often affects those older than 65 years). However, influenza A has a substantial health effect on every age group.

Due to the limited therapeutic options for influenza and significant morbidity and mortality despite treatment, additional therapeutics are warranted. One potential therapeutic that is fairly rapidly available is the use of anti-influenza A immune plasma as immunotherapy.

The objective of this protocol is collection of anti-influenza A immune plasma from male volunteers that meet criteria for use in human plasma therapy studies. The use of plasma from male donors will minimize the risk of transfusion related acute lung injury (TRALI), which has been associated with antibodies (likely generated during pregnancy) found in female plasma. For this reason, only male donors will be enrolled.

This protocol does not administer any investigational product, but rather collects plasma from subjects with a high anti-influenza A antibody titer (convalescent survivors of influenza infection or recipients of a licensed influenza vaccine).

Following screening of potential subjects to identify those who are not eligible to participate in plasma donations and to determine the likelihood of having antibodies to influenza A (H1N1 or H3N2) from a recent infection or immunization, enrolled subjects will receive a baseline physical and laboratory examination. Eligible subjects with high influenza A hemagglutination inhibition (HAI) titers will then be scheduled for at least 3 (and up to 20) plasma collection sessions. Following testing of the collected plasma for potential pathogens, it may be used as therapeutic plasma, and/or it may be used for the manufacturing of high titer anti-influenza A intravenous immune globulin (IVIG). Both options would support clinical trials aimed at developing additional therapeutics for influenza infection.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Provide written informed consent before initiation of any study procedures.
  2. Male adults between the ages of 18 and 60 years old
  3. History suggestive of having anti-influenza A antibodies (either of the following):

     1. An influenza like illness (e.g. fever, chills, malaise, cough, myalgias and nausea) consistent with influenza A infection. Subjects must not be symptomatic and be at least 7 days since the resolution of fever, and must enroll within 12 months of illness.
     2. Vaccination with a licensed influenza vaccine and at least 14 days following the last vaccination in the series, and enrolling within 12 months of vaccination.
     3. Some subjects may meet both requirements and enrollment should be within 12 months of the most recent event (illness or vaccination)
  4. Adequate clinical parameters (all of the following):

     1. Afebrile (temperature < 38 Degrees C)
     2. Systolic blood pressure > 100 and < 180 mmHg
     3. Diastolic blood pressure > 50 and < 100 mmHg
     4. Heart rate between 50-100 beats/minute (Individual site blood establishment's SOPs may also permit healthy athletic subjects with heart rates < 50 beats/minutes to donate plasma, and, if so, subjects with heart rates < 50 beats/minutes may participate in this study)
  5. Weight greater than or equal to 110 pounds (50 kg)
  6. Adequate peripheral venous access for plasma donation (as judged by the examiner)
  7. Willingness to have samples stored

     EXCLUSION CRITERIA:

  <!-- -->

  1. Any sign of active influenza, (as judged by the investigator) including but not limited to:

     1. Subjective or documented fever (> 38 Degrees C)
     2. Cough
     3. Shortness of breath
     4. Diarrhea
  2. Has a medical history of

     1. Thrombocytopenia or other blood dyscrasias
     2. Congestive heart failure
     3. Pulmonary hypertension
     4. Bleeding diathesis or therapeutic anticoagulation
     5. Human immunodeficiency virus (HIV)/AIDS
     6. Hepatitis B
     7. Hepatitis C
     8. Known history of hepatitis after the 11th birthday
     9. Trypanosomiasis (Chagas' disease and sleeping sickness)
     10. Leishmaniasis (Kala-azar)
     11. Filariasis
     12. Q fever
     13. Yaws
  3. History of cancer that meets any one of the following criteria:

     1. Leukemia or lymphoma: permanent deferral
     2. Melanoma: 10 year deferral (with exception of melanoma-in-situ: defer until biopsy site is healed)
     3. Squamous cell or basal cell cancer of skin: defer until excision site is healed
     4. All other cancers: defer for 2 years since end of treatment
  4. Medication history that includes any of the following:

     1. Current use of oral or parenteral steroids, high-dose inhaled steroids (> 800 μg/day of beclomethasone dipropionate or equivalent) or other immunosuppressive or cytotoxic drugs
     2. Finasteride (Proscar, Propecia) within the last 1 month
     3. Isotretinoin (Accutane) within the last 1 month
     4. Acitretin (Soriatane) within the last 3 years
     5. Etretinate (Tegison) at any time
     6. Dutasteride (Avodart) within the last 6 months
     7. Growth hormone made from human pituitary glands at any time
     8. Beef insulin from the United Kingdom at any time
     9. Warfarin (Coumadin) within the last 1 week
     10. Antibiotics within the prior 48 hours
  5. Has ever had any of the following:

     1. Sexual contact with someone known to have HIV
     2. Had a relative with Creutzfeldt-Jakob Disease, or been told that this disease is inherited within the family
     3. Received blood transfusion in the United Kingdom
     4. History of receiving money, drugs or other payment for sex
     5. History of receiving clotting factor concentrates
     6. History of a dura mater graft
     7. History of babesiosis
     8. For male donors, history of sexual contact with another male
     9. Used needles to take drugs, steroids, or other medications not prescribed by a physician
     10. Was born, lived in, had blood donation in or ever had sexual contact with anyone who lived in Cameroon, Central African Republic, Chad, Congo, Equatorial Guinea, Gabon, Niger, or Nigeria after 1977
     11. History of living 3 or more months total (need not be consecutive) in the UK from 1980-1996
     12. History of living 5 or more years total (need not be consecutive) in Europe since 1980
     13. History of living 6 or more months total (need not be consecutive) on a U.S. military base in Europe from 1980-1996 (specifically from 1980 through 1990 in Belgium, the Netherlands, or Germany, and from 1980 through 1996 in Spain, Portugal, Italy, or Greece)
  6. Within the 8 weeks prior to enrollment:

     a. Was vaccinated with the small pox vaccine, or was in close contact with someone who was vaccinated (i.e., close family member)
  7. Within the 4 months prior to enrollment has had:

     a. A blood donation of a double unit of red cells
  8. Within the 12 months prior to enrollment has:

     1. Received any blood or blood component
     2. Donated blood at a paid donation center (donations at a hospital blood establishment do not apply)
     3. History of tattoo application
     4. History of unsafe (multiple-use equipment) acupuncture, or piercing practices
     5. Received an organ transplant
     6. Received a bone or skin graft
     7. Lived with someone who has any type of hepatitis
     8. Been incarcerated for more than 72 hours
     9. Oral or inhalation use of illegal drugs (i.e., those not prescribed by a physician)
     10. Had or has been treated (with or without confirmatory diagnosis) for syphilis or gonorrhea
  9. Within the last 12 months has had sexual contact with (any of the following):

     1. An individual having viral hepatitis
     2. A prostitute or anyone else who takes money or drugs or other payment for sex
     3. Anyone who has ever used needles to take drugs, steroids, or anything else not prescribed by their doctor
     4. Anyone who has hemophilia or has used clotting factor concentrates
     5. For females, a male who has ever had sexual contact with another male
  10. Participation in medical research that includes:

      1. Protocols that are currently ongoing or will start during the duration of this study that require more than 100 mL of blood to be given in any 8-week period of time
      2. Administration of any unlicensed drug within the last 3 months or during the duration of this study
      3. Administration of any unlicensed vaccine within the last 12 months or during the duration of this study.
  11. Subjects that have participated in previous plasma collection or other cell component collection within the last 3 months may have restrictions to participation based on the site plasma collection SOP. In this scenario, discussion should occur with the blood establishment to ensure eligibility to donate plasma.

PLASMA DONATION CRITERIA (all of the following):

1. Anti-Influenza A HAI titer of 1:160 or greater and H3N2 HAI titer of at least 1:40
2. Adequate laboratory parameters from screening (must meet all of the criteria below)

   1. Hemoglobin level of greater than or equal to 12.5 g/dL
   2. HCT greater than or equal to 38%
   3. Platelets greater than or equal to 150 x 10^3/cubic mm
   4. Total serum protein greater than or equal to 6.0 g/dl
   5. Quantitative immune globulin levels (all of the following)

      1. Ig A greater than or equal to 90 mg/dL
      2. Ig G greater than or equal 650 mg/dL
      3. Ig M greater than or equal 35 mg/dL
   6. Review of other screening labs should ensure no other underlying medical condition that would increase subject's risk of apheresis.
3. Negative serologic and molecular tests for blood borne pathogens, to include:

   1. Anti-HIV-1/2
   2. Anti-HTLV-I/II
   3. Anti-HCV
   4. HBsAg (hepatitis B surface antigen)
   5. Serologic test for syphilis (PK-TP)
   6. HIV NAT
   7. HCV NAT
   8. WNV NAT

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Male subjects with a history consistent with influenza infection and/or vaccination against influenza.
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2009-09; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Collection of Anti-Influenza A Immune Plasma | Individual duration is a maximum of 240 days per subject.
  Subjects will be scheduled for at least 3, and up to 20, plasma collection procedures.

CONTACTS AND LOCATIONS:
Locations (12):
- United States (12):
  - UCLA Care Center, Los Angeles, California
  - UCLA Pediatric Infectious Diseases, Los Angeles, California
  - University of Colorado Hospital Blood Donor Center, Aurora, Colorado
  - Rush University Medical Center, Chicago, Illinois
  - Johns Hopkins University, Baltimore, Maryland
  - National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland
  - AIDS Clinical Trials Unit, NYU School of Medicine, New York, New York
  - Cornell Clinical Trials Unit, New York Presbyterian Hospital, Weill Cornell Medical College, New York, New York
  - Clinical Translational Research Center (CTRC) at UNC Hospitals, Chapel Hill, North Carolina
  - AIDS Clinical Trial Unit, Holmes Hospital, Div of Infectious Disease, University of Cincinnati College of Medicine, Cincinnati, Ohio
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Washington, Seattle, Washington

REFERENCES:
- [Background] Morse SS. Factors in the emergence of infectious diseases. Emerg Infect Dis. 1995 Jan-Mar;1(1):7-15. doi: 10.3201/eid0101.950102. PMID 8903148
- [Background] Bean WJ, Schell M, Katz J, Kawaoka Y, Naeve C, Gorman O, Webster RG. Evolution of the H3 influenza virus hemagglutinin from human and nonhuman hosts. J Virol. 1992 Feb;66(2):1129-38. doi: 10.1128/JVI.66.2.1129-1138.1992. PMID 1731092
- [Background] de Jong MD, Tran TT, Truong HK, Vo MH, Smith GJ, Nguyen VC, Bach VC, Phan TQ, Do QH, Guan Y, Peiris JS, Tran TH, Farrar J. Oseltamivir resistance during treatment of influenza A (H5N1) infection. N Engl J Med. 2005 Dec 22;353(25):2667-72. doi: 10.1056/NEJMoa054512. PMID 16371632
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/detail/A_2009-I-0226.html